CLINICAL TRIAL: NCT01529437
Title: Phase 1 Single Center, Randomized, Controlled Study Using Sublingual Immunotherapy for Timothy Grass and Dust Mite Allergies
Brief Title: Sublingual Immunotherapy Studies for Grass and Dust Mite Allergies
Acronym: SLIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kari Christine Nadeau, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8669
Record Dates: First submitted 2012-01-30; First posted 2012-02-08 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Allergies; Allergic Rhinitis; Asthma
Keywords: allergy; immunology; immune tolerance; immunotherapy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic; Asthma | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sublingual immunotherapy (Active Comparator): Subjects will take sublingual immunotherapy who have dust mite and timothy grass allergies
  Interventions: Drug: sublingual immunotherapy
- placebo arm (Placebo Comparator): The placebo arm will be double blinded and is an important control in SLIT therapies
  Interventions: Drug: sublingual immunotherapy; Drug: placebo sublingual immunotherapy

INTERVENTIONS:
Drug: sublingual immunotherapy — Sublingual immunotherapy is provided in an extract form under IND 13485 and dosed safely through a maintenance dose of 12 months.
Drug: placebo sublingual immunotherapy — SLIT placebo will be the same color and consistency of the active drug arm to provide double blinding
  Arms: placebo arm

SUMMARY:
This is a study for children and adults who are interested in a new therapy for their allergies to dust mite and timothy grass. The new therapy is called sublingual immunotherapy and the investigators are testing if it is safe and well tolerated.

DETAILED DESCRIPTION:
This is a phase I, single-center, randomized, placebo-controlled study of sublingual immunotherapy (SLIT) in pediatric and adult subjects with both house dust mite (HDM) and timothy grass (TG) allergies. We will evaluate whether Dermatophagoides farinae (DF) and/or TG allergen SLIT is safe in children and adults. We will also determine whether treatment with DF and/or TG SLIT reduces the severity of allergic symptoms (allergic rhinitis, allergic conjunctivitis) and enhances their resolution. The study will also evaluate whether SLIT provides a robust durability of response once it is terminated. The dosing-phase of the study will last up to 12 months. In addition, a follow up period of 2 years will occur. Approximately 10 subjects will be on placebo, and 20 on active treatment.

ELIGIBILITY:
SUBJECT INCLUSION CRITERIA:

1. Pediatric and adult timothy grass- and Dermatophagoides farinae-sensitive subjects with allergic rhinoconjunctivitis with or without asthma perennially or during grass pollen season.
2. Subjects must be 5 years of age or older.
3. Sensitivity to the relevant allergen will be documented by a positive skin prick test result (see Appendix E for details).
4. All female subjects of child-bearing potential will be required to provide a urine sample for pregnancy testing that must be negative one week before being allowed to participate in the study.
5. Subjects must be planning to remain in the study area during the trial.
6. Subjects and/or their parents must be trained on the proper use of the Epi-Pen to be allowed to enroll in the study.
7. Subjects and/or their parents must be mentally and physically capable of self-administering oral drug.

SUBJECT EXCLUSION CRITERIA:

No absolute contraindications to allergen skin testing and/or sublingual immunotherapy are known. However, the risk of serious systemic anaphylactic reactions to pollen or any potent allergenic extract suggests a number of preexisting conditions that should be considered relative contraindications. Among those conditions are acute infections, autoimmune disease, severe cardiac disease, and treatment with beta-adrenergic antagonistic drugs (beta-blockers).

1. Subjects having a history of unexplained anaphylaxis within 2 years or a history of multiple (≥2) episodes of anaphylaxis in the past year, frequent allergic or non-allergic urticaria, or history consistent with poorly controlled persistent asthma. Anaphylaxis must be medically diagnosed.
2. Subjects with unstable angina, significant arrhythmia, uncontrolled hypertension, chronic sinusitis, or other chronic or immunological diseases that in the mind of the investigator might interfere with the evaluation or administration of the test drug or pose additional risk to the subject e.g. gastrointestinal or gastroesophageal disease, chronic infections, scleroderma, hepatic and gallbladder disease, chronic non-allergic pulmonary disease.
3. Subject with an FEV1 or PEF less than 80% predicted (moderate persistent asthma) with or without controller medication.
4. Subjects who have received an experimental drug in the last 30 days prior to admission into this study or who plan to use an experimental drug during the study.
5. Subjects who have received timothy grass or dust mite allergen immunotherapy within 3 years prior to admission in this study.
6. Subjects who are current users of oral, intramuscular, or intravenous corticosteroids, tricyclic antidepressants, or are taking a beta-blocker (oral or topical).
7. Subjects routinely using medication that could induce adverse gastrointestinal reactions during the study.
8. Subjects refusing to sign the EpiPen Training Form (see Appendix F).
9. Pregnant or breast feeding females.
10. Subjects who have any symptoms at dose levels 1 or 2 at the Preliminary Dosing Visit (see, below).
11. Subjects with significant pet allergies who have significant exposure at home or at work.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome is safety | 2008-2014 (6 years)
  We will assess safety outcomes according to GCP/CFR and NIAID guidelines
The number of adverse events in the placebo vs the treatment arm will be compared | 2008-2016
  Adverse events will be defined by GCP/CFR and by NIAID guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nadeau, MD, PhD, Principal Investigator — Stanford University Faculty
Locations (1):
- Stanford University, Stanford, California, United States